CLINICAL TRIAL: NCT02732847
Title: Post-Dated Versus Voluntary Delayed Antibiotic Prescriptions for Acute Respiratory Infections in Primary Care: A Randomized Trial
Brief Title: Trial of Post-Dated Delayed Antibiotic Prescriptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: worrall1
Record Dates: First submitted 2010-05-27; First posted 2016-04-11 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2006-06

CONDITIONS: Acute Upper Respiratory Tract Infections
Keywords: Respiratory infections; Primary care; Antibiotics; Delayed prescriptions
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post-Dated Prescription (Other): a delayed prescription dated 2 days after clinical office visit
  Interventions: Other: A delayed prescription dated 2 days after clinical office visit
- Usual (Other): usual date
  Interventions: Drug: Usual Dated

INTERVENTIONS:
Other: A delayed prescription dated 2 days after clinical office visit
  Arms: Post-Dated Prescription
Drug: Usual Dated
  Arms: Usual

SUMMARY:
Delayed prescriptions have been shown to lower antibiotic use for upper respiratory tract infections (which are mostly viral).

This trial will test the hypothesis that if the clinician post-dates the delayed prescription by 2 days, rather than dating it on the day the patient is seen, there will be a further drop in the rate of antibiotic use.

DETAILED DESCRIPTION:
6 family doctors and 2 nurse practitioners in a small rural town will issue delayed antibiotic prescriptions to adult patients with new acute respiratory tract infections. The delayed prescriptions will be randomly dated for either the day of the office visit, or 2 days later. The 2 local pharmacies will note whether the prescription is cashed, and when.

It is hypothesised that post-dating the prescription will result in a reduced cashing rate.

Each arm of the study (Usual v Post-Dated) will contain 75 subjects. This sample will have the power to detect a 25% change in prescription use.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Adults with an untreated upper respiratory tract infection
* Adults presenting for the first time to a family physician or a nurse practitioner

Exclusion Criteria:

* Less that 18 years
* Having a clear indication for antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial University, St. John's, Newfoundland and Labrador, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual: usual date
  Usual Dated
Period: Overall Study
Arm/Group | Post-Dated Prescription | Usual
Started | 75 | 74
Completed | 33 | 32
Not Completed | 42 | 42
Not completed — some filled early | 42 | 42

BASELINE CHARACTERISTICS:
Population: This was an ad hoc study, and therefore no baseline information was recorded for this study design
Groups:
- Total: Total of all reporting groups
Arm/Group | Post-Dated Prescription | Usual | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Filled a Prescription in 20 Days
Description: Prescriptions
Time Frame: 20 days
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Dated Prescription | Usual
Number analyzed (Participants) | 33 | 32
Participants | 16 | 16
Statistical Analysis 1: Comparison: Post-Dated Prescription vs Usual; Test type: Other — Chi square tests used to compared groups; p = 0.924, Chi-squared — A p-value of < 0.05 was considered

ADVERSE EVENTS:
Time Frame: This study did not involve reporting of adverse reactions over the 19 days time span
Description: This study was educational in nature. It was designed to just determine the timing of the number of the prescriptions filled by individuals. It is did not involve the gathering of any information on adverse effects.
Arm/Group | Post-Dated Prescription | Usual
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No